CLINICAL TRIAL: NCT00292422
Title: A Randomized, Blinded, Placebo-Controlled, Multicenter, Dose-Escalating Study to Evaluate the Safety, Tolerability and Pharmacokinetics of BG9924 When Given in Combination With Methotrexate to Subjects With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to DMARD Therapy
Brief Title: Dose-Escalating Study of BG9924 in Combination With Methotrexate in Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec Medical Director, Biogen Idec Inc.
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 104-RA-201
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2007-12-31 (Estimated); Status verified 2007-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis, Rheumatoid; Methotrexate; Antirheumatic Agents
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: BG9924

SUMMARY:
This Phase 2a study is designed to evaluate the safety and tolerability of multiple subcutaneous (SC) doses of BG9924, administered in a cohort dose-escalation fashion, in patients with active rheumatoid arthritis (RA) who have had an inadequate response to therapy with disease-modifying anti rheumatic drugs (DMARDs) and who may have undergone anti-TNF therapy. This study will assist with dose selection for further planned Phase 2 studies.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent. If required by local law, candidates must also authorize the release and use of protected health information (PHI).
* Male or female subjects aged 18 to 75 years old, inclusive, at the time informed consent is given.
* Must have a diagnosis of RA Functional Class I-III according to the 1987 Revised American Rheumatism Association Criteria for the Classification of Rheumatoid Arthritis for at least 6 months prior to baseline.
* Must have been treated with MTX (>=10 mg/week to <=25 mg/week) for at least 3 months immediately prior to enrollment. The dose of MTX must be stable for at least 4 weeks prior to Day 0.
* Must have active disease at Screening defined as SJC >=5 (66 joint count) and TJC >=5 (68 joint count).
* All DMARDs, other than MTX or hydroxychloroquine sulfate, must be withdrawn at least 4 weeks prior to Day 0 (8 weeks for infliximab, adalimumab, and leflunomide).
* Male and female subjects of child-bearing potential must be willing to practice effective birth control for the duration of the study. Female subjects must be: (1) postmenopausal for at least 12 months, (2) surgically sterile, or (3) willing to use 2 documented forms of birth control (e.g., barrier and spermicide, intrauterine device and barrier or spermicide, or birth control pill and barrier or spermicide).
* Subjects must be willing and able to complete all planned study procedures.

Exclusion Criteria:

* Subjects with a history of a malignancy or carcinoma in situ (subjects with a history of excised or treated basal cell carcinoma are eligible to participate in this study).
* Moles or lesions currently undiagnosed, but suspicious for malignancy.
* Subjects with a history of clinically significant (as determined by the Investigator) cardiac, allergic, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal or hematologic insufficiency or major disease.
* Subjects with rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA (including but not limited to vasculitis, pulmonary fibrosis or Felty's syndrome). Secondary Sjögren's syndrome is permitted.
* Serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, septicemia) within 3 months prior to Day 0.
* History of recurrent significant infections.
* Primary or secondary immunodeficiency (history of or currently active).
* History of tuberculosis or positive purified protein derivative (PPD; positive Mantoux test defined as ³10 mm of induration [size of raised bump, not redness]) test during the screening period. Subjects whose PPD induration is >=5 mm but <10 mm are eligible for the study if they have a negative chest X-ray during the screening period.
* Fever (body temperature >38°C) or symptomatic viral infection or bacterial infection within 2 weeks prior to Day 0.
* Receipt of live vaccine within 4 weeks prior to Day 0.
* Clinically significant chest X-ray abnormality within 3 months prior to Screening.
* Current or prior treatment with more than 1 anti-TNF agent (etanercept, infliximab, or adalimumab) or other approved or investigational biologic agent for the treatment of RA.
* Previous treatment with an anti-a4 integrin antibody within the last 6 months.
* Anti-TNF therapy with infliximab or adalimumab within 8 weeks or etanercept within 4 weeks prior to Day 0.
* Treatment with another investigational drug within the 3 months prior to Day 0 or within 5 half-lives of the agent, which ever is longer.
* If the subject has previously received cell-depleting therapies, relevant cell counts must have returned to normal.
* Subjects will be excluded who meet any of the following criteria regarding treatment with concomitant therapy for RA:

  * Concomitant use of an oral steroid exceeding 10 mg/day of prednisone (or equivalent dose) or, if 10 mg/day or less, was not administered at a stable dose for at least 4 weeks prior to Day 0.
  * Concomitant use of an NSAID that was not administered at a stable dose for at least 2 weeks prior to Day 0.
  * Concomitant use of hydroxychloroquine sulfate at >400 mg/day or not administered at a stable dose for 4 weeks prior to Day 0.
  * Concomitant use of other anti-arthritic treatments, including approved or experimental oral or topical agents, within 4 weeks prior to Day 0.
  * Intra-articular corticosteroid injections within 4 weeks prior to Day 0.
  * Previous exposure to BG9924.
* Subjects will be excluded who underwent any surgical procedure, including bone/joint surgery/synovectomy (including joint fusion or replacement), within 12 weeks prior to baseline or who are planning such a procedure within 16 weeks after randomization.
* Subjects with any laboratory test result at Screening considered clinically significant (as determined by the Investigator) or

  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times the upper limit of normal (ULN) established by the central laboratory
  * Platelet count <150,000/μL
  * Hemoglobin <8.5 g/dL
  * Neutrophil count <1.5-10^3/μL
* Positive for hepatitis C virus (HCV), hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV; it is recognized that HIV testing may not be permitted at all sites).
* Nursing mother, pregnant women and women who are planning to become pregnant while in the study.
* Blood donation (1 unit or more) within 1 month prior to screening.
* History of drug or alcohol abuse (as determined by the Investigator) within 1 year prior to Day 0.
* Current enrollment in any other investigational drug study.
* Previous participation in this study.
* Subjects who are expected to be unavailable for the duration of the trial, likely to be noncompliant with the protocol, or who are felt to be unsuitable by the Investigator/Sponsor for any other reason.
* Other unspecified reasons that, in the opinion of the Investigator/Sponsor, make the subject unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of BG9924 when administered in combination with MTX to subjects with active RA who have had an inadequate response to DMARD therapy

SECONDARY OUTCOMES:
To assess the pharmacokinetics and pharmacodynamics of multiple doses of BG9924 in this patient population
To assess the preliminary efficacy of multiple doses of BG9924 in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Evan Beckman, MD, Study Director — Biogen
Locations (10):
- United States (3):
  - Fiechtner Research Inc., Lansing, Michigan
  - Arthritis Consultants Inc., St Louis, Missouri
  - The Arthritis Group, Philadelphia, Pennsylvania
- Poland (7):
  - Centrum Medyczne SpecjalistycznyGabinet Lekarski, Bialystok
  - Oddzial Reumatologii Wojewodzki Szpital, Elblag
  - Osrodek Badan Klinicznych, Lublin
  - Prakyta Lekarza Rodzinnego "Nasz Lekarz", Torun
  - Klinika Chorob Tkanki Lacznej-Instytut Reumatologiczny, Warsaw
  - Klinika Reumatologii-Instytut Reumatologiczny, Warsaw
  - Centrum Leczenia Chorob Cywilizacyjnych, Warsaw